CLINICAL TRIAL: NCT02163369
Title: The Use of Aromatherapy for Symptom Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central DuPage Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-031-1
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Nausea, Vomiting and Anxiety Associated With Medical Oncology Patients
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peppermint and Lavender Essential Oils (Experimental)
  Interventions: Drug: Peppermint and Lavender Essential Oils

INTERVENTIONS:
Drug: Peppermint and Lavender Essential Oils

SUMMARY:
The purpose of this pilot study is to introduce the use of aromatherapy/essential oils to medical oncology patients at Central DuPage Hospital to assess their perceived effectiveness to relieve symptoms of nausea or vomiting and/or anxiety.

Peppermint oil will be used for nausea/vomiting and lavender oil will be used for anxiety. This study will involve administration of aromatherapy to a convenience sample of patients, who will then be asked to complete a brief questionnaire. The questionnaire will involve a simple likert scale to measure efficacy (in the opinion of the patient) and simple multiple-choice questions to determine patients' likeliness to use aromatherapy again.

ELIGIBILITY:
Inclusion Criteria:

* Adult hospitalized medical oncology patients admitted to Central DuPage Hospital.
* Age 18 years or greater.
* Able to understand and speak English.
* Women of non-childbearing potential or with childbearing potential with a negative pregnancy test documented during the hospital stay.
* Able to understand concept of aromatherapy for treatment of distressing symptoms.

Exclusion Criteria:

* Prisoners.
* Non-English speaking patients.
* Under the age of 18.
* Unable to comprehend the concept of aromatherapy.
* Severe cognitive impairment.
* Not experiencing the symptoms of nausea, vomiting or anxiety.
* Women with child-bearing potential who have not had a negative pregnancy test during the hospital stay.
* Patients with known allergy to lavender or peppermint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Post Intervention Patient Interview Form | 24hrs post aromatherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lyons, MSN, APN/CNS, RN-BC, ONC, Principal Investigator — Central DuPage Hospital
Locations (1):
- Central DuPage Hospital, Winfield, Illinois, United States